CLINICAL TRIAL: NCT07246226
Title: Communication in the Surgical Environment to Promote a Climate of Safety: Implementation of Evidence
Brief Title: Communication in the Surgical Environment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cintia Silva Fassarella (Other)
Responsible Party: Sponsor-Investigator, Cintia Silva Fassarella, Doctor, Rio de Janeiro State University
Organization: Rio de Janeiro State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 7.924.577
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Communication in the Surgical Environment
Keywords: Organizational Culture; Implementation Science; Patient Safety; Surgicenters; Patient Care Team

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- surgical team (Other): Participants will complete an audit questionnaire before and after the implementation of the surgical briefing protocol.
  Interventions: Behavioral: Surgical communication training

INTERVENTIONS:
Behavioral: Surgical communication training — Seminar on communication in the surgical environment with lectures and training on how to conduct surgical briefings

SUMMARY:
The objective of this evidence implementation is to identify whether the implementation of a surgical briefing protocol promotes the strengthening of communication in the surgical environment of safety in the operating room among the orthopedic surgery team, including nurses, nursing technicians, orthopedic surgeons, and anesthesiologists.

The main question it seeks to answer is: does the surgical briefing protocol used to promote the strengthening of communication in the surgical environment and safety culture in the operating room comply with best practices? Participants will be asked to complete a baseline audit questionnaire, participate in training on the implementation of the surgical briefing protocol, and subsequently complete a follow-up audit questionnaire.

DETAILED DESCRIPTION:
The aim of the study is to identify whether the implementation of a surgical briefing protocol promotes the strengthening of the 'communication in the surgical environment' domain of safety climate in the operating room. A multi-method study is proposed to be developed in the surgical center of a university hospital located in the city of Rio de Janeiro. The study will be carried out in two phases: In Phase I, a surgical briefing protocol will be developed, validated and implemented that will follow the JBI (Joanna Briggs Institute) methodology of evidence implementation. As a support for methodological rigor, the tool SQUIRE2.0 (Standards for QUalityImprovement Reporting Excellence): revised publication guidelines from a detailed consensus process will be used. Finally, Phase II will have a quantitative approach with a cross-sectional design, using the Safety Attitudes Questionnaire/Operating Room (SAQ/OR). As a support for methodological rigor, the tool Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) will be used. The population will be composed of: nurses, nursing technicians, surgeons and anesthesiologists who work in orthopedic surgery and management of the unit. Regarding sampling, for Phase I of the study, a focus group will be constituted, called a working group (WG), adopting an intentional sampling, ensuring the participation of all health professional categories that work in orthopedic surgery. The inclusion criteria will be health professionals who work at least 20 hours per week, working in orthopedic surgeries and/or managers of the surgical center. For the validation stage, professionals withhigher education with specialization in the operating room (for nursing professionals) or orthopedic surgery (for medical professionals) will be adopted as inclusion criteria, as well as professors and researchers whose lines of research are directly related to surgical communication, patient safety and safety culture. For Phase II, a non-probabilistic sampling will be adopted, the sample calculation will be performed with the aid of the EpiInfo v5.5.9 application, adopting a confidence level of 95%. For this sample, health professionals who work at least 20 hours a week, who work directly or indirectly in patient care and who have been working in the sector for at least one month will be adopted as inclusion criteria. The exclusion criteria were the professionals who will compose the focus group. It is expected to implement a surgical briefing protocol and advance in the implementation of evidence to promote the maturation of the safety culture in the operating room, fostering safer surgical care, especially in this highly specialized sector that is the operating room. In addition to encouraging future studies involving the science of implementation in safety culture, allowing research to be truly focused on the best available evidence. It is intended that the research serves as a source of data on patient safety in the surgical environment and offers an innovative model to evaluate and intervene in complex aspects of the safety culture, involving professionals and senior management in health in the surgical environment.

ELIGIBILITY:
Inclusion Criteria: healthcare professionals who work at least 20 hours per week, directly or indirectly involved in patient care -

Exclusion Criteria: professionals with less than 30 days of experience in the sector

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of improved safety climate in the operating room | From the registration period until the end of the protocol implementation, in 4 months
  Quantitative data will be manually entered into a spreadsheet (Microsoft Excel®) and subsequently imported into the R program, version 4.2.1. The analysis will be performed using descriptive statistics (absolute and relative frequency) and mean and standard deviation. Blank items and "not applicable" items will be excluded from the analysis, as will questionnaires with the same answer to all questions. An improvement is considered if the mean is 75 or higher.

CONTACTS AND LOCATIONS:
Locations (1):
- UERJ, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No